**Document Date:** April 7, 2020

EFFECT OF EXPIRATORY MUSCLE TRAINING ON STOMATOGNATHIC SYSTEM

IN PATIENTS WITH STROKE

Ömer DURSUN PT, PhD1. Tamer ÇANKAYA, PT, Assoc. Prof. Dr2. Erdal DİLEKÇİ, MD,

Assoc. Prof. Dr<sup>3</sup>.

**Statistical Analysis** 

SPSS 22.0 was used for the data analysis. While constant variables were given as mean  $\pm$  standard

deviation, categoric variables were given as number and percentage. If the parametric test conjectures

were ensured, materiality test between two means was used for independent group variable

comparison. If the parametric test conjectures were not ensured Mann-Whitney U test was used for

independent group variable comparison. In dependent group analyses, materiality test was used

between two couples in case parametric test conjectures were ensured, if the parametric test

conjectures were not ensured Wilcoxon test was used.